CLINICAL TRIAL: NCT01704235
Title: Community Based Participatory Research to Understanding Symptom Perception, Preventive Care-Seeking, and Their Impact on Cervical Cancer Screening Among Vietnamese American Women
Brief Title: Vietnamese Women's Health Project III
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00008709; CPC-12122-L (Other: OHSU)
Record Dates: First submitted 2012-10-04; First posted 2012-10-11 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Cervical Cancer
Keywords: screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary health care providers: medical physicians and nurse practitioners
  Interventions: Other: Demographic Form and Semi-Structured Interview Guide

INTERVENTIONS:
Other: Demographic Form and Semi-Structured Interview Guide — The demographic form will include the following items: age, age at immigration, years lived in the United States, Vietnamese speaking ability, and marital status. In addition for participants who are primary health care providers, the following items will be included: annual income before taxes, gender, race and ethnicity, specialty area of practice, and number of years practicing as a primary health care provider, practice setting, and country received Pap test training.
  A semi-structured interview guide will also be used and will include possible probing questions. A semi-structured interview guide was developed with the research team.

SUMMARY:
The purpose of this protocol is to understand the extent of symptom perception and preventive care-seeking among Vietnamese American women and their impact on cervical cancer screening from the perspectives and experiences of key informants including primary health care providers and Vietnamese American women (VAW, foreign-born and United States-born). With this information, the investigators can better understand how to promote cervical cancer screening in the Vietnamese community.

DETAILED DESCRIPTION:
No further extensive description.

ELIGIBILITY:
Inclusion Criteria:

* Primary health care providers are eligible to participate in the study if they meet the following criteria:

  * self-identify as currently practicing as a primary licensed independent practitioner including as a medical physician or nurse practitioner,
  * whose service populations include Vietnamese American women,
  * and are able to understand and speak English or Vietnamese.
* Vietnamese American women are eligible to participate in the study if they meet the following criteria:

  * self-identify as a Vietnamese American woman (foreign-born women who have immigrated to the United States from other countries or are United States-born),
  * between ages 21 to 65 years old,
  * have not had a hysterectomy,
  * and are able to understand and speak English or Vietnamese.

Exclusion Criteria:

* Not a Vietnamese American woman
* Not between the ages of 21 to 65 years old
* Had a hysterectomy

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential participants will be recruited from the Portland, Oregon Metropolitan area through referrals and snowball method. Primary health care providers are eligible to participate in the study if they meet the following criteria: self-identify as currently practicing as a primary licensed independent practitioner including as a medical physician or nurse practitioner, whose service populations include Vietnamese American women, and are able to understand and speak English or Vietnamese. Vietnamese American women are eligible to participate in the study if they meet the following criteria: self-identify as a Vietnamese American woman, between ages 21 to 65 years old, have not had a hysterectomy, and are able to understand and speak English or Vietnamese.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2016-07-25 (Actual)

PRIMARY OUTCOMES:
The extent of symptom perception | Duration of the study; Up to 1 year
  To understand the extent of symptom perception among Vietnamese American women (foreign and United States-born) and their impact on cervical cancer screening from the perspective and experiences of key informants including primary health care providers. A semi-structured interview guide will be used to assess the extent of preventive care-seeking. The interview guide includes the following topics: thoughts and experiences regarding Vietnamese American women's knowledge and beliefs about how cervical cancer develops, thoughts and experiences regarding Vietnamese American women and use of cancer screening tests such as cervical cancer screening for early detection/preventive health care, thoughts and experiences about Vietnamese American women's lack of familiarity with the term Pap smear or a Pap test, and thoughts and experiences regarding Vietnamese American women's decision and timing to seek medical care and preventive health care.

SECONDARY OUTCOMES:
The extent of preventive care-seeking | Duration of the study; Up to 1 year
  To understand the extent of preventive care-seeking among Vietnamese American women (foreign and United States-born) and their impact on cervical cancer screening from the perspective and experiences of key informants including primary health care providers. A semi-structured interview guide will be used to assess the extent of preventive care-seeking. The interview guide includes the following topics: thoughts and experiences regarding Vietnamese American women's knowledge and beliefs about how cervical cancer develops, thoughts and experiences regarding Vietnamese American women and use of cancer screening tests such as cervical cancer screening for early detection/preventive health care, thoughts and experiences about Vietnamese American women's lack of familiarity with the term Pap smear or a Pap test, and thoughts and experiences regarding Vietnamese American women's decision and timing to seek medical care and preventive health care.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Nail, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States